CLINICAL TRIAL: NCT03965234
Title: Phase I/ II Study of Pulmonary Suffusion to Control Minimal Residual Disease in Resectable or Ablatable Sarcoma or Colorectal Pulmonary Metastases
Brief Title: Pulmonary Suffusion in Controlling Minimal Residual Disease in Patients With Sarcoma or Colorectal Metastases
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: i 70818; NCI-2019-02940 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); i 70818 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2019-05-22; First posted 2019-05-28 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Bone Sarcoma; Metastatic Malignant Neoplasm in the Lung; Metastatic Soft Tissue Sarcoma; Metastatic Unresectable Sarcoma; Resectable Sarcoma; Colorectal Cancer
MeSH Terms: conditions — Bone Neoplasms; Sarcoma; Colorectal Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Metastasectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Prevention (cisplatin, metastasectomy) (Experimental): Patients undergo pulmonary suffusion consisting of cisplatin via infusion. Patients the undergo metastasectomy. Beginning 4-8 weeks, patients with unresectable sarcoma may receive chemotherapy.
  Interventions: Drug: Cisplatin; Procedure: Isolated Chemotherapeutic Lung Perfusion; Procedure: Metastasectomy

INTERVENTIONS:
Drug: Cisplatin — Given via infusion
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Isolated Chemotherapeutic Lung Perfusion — Undergo pulmonary suffusion
  Other Names: isolated lung perfusion
Procedure: Metastasectomy — Undergo metastasectomy

SUMMARY:
This phase I/II trial studies the side effects of pulmonary suffusion in controlling minimal residual disease in patients with sarcoma or colorectal carcinoma that has spread to the lungs. Pulmonary suffusion is a minimally invasive delivery of chemotherapeutic agents like cisplatin to lung tissues. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Pulmonary suffusion may also be useful in avoiding later use of drugs by vein that demonstrate no effect on tumors when delivered locally.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of chemotherapy isolated to the pulmonary circulation by determining the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) of each chemotherapy agent. (Phase I) II. To determine the rate of local recurrences in patients receiving pulmonary suffusion, compared to historical controls in patients with completely resected pulmonary metastases (unilateral and bilateral disease). (Phase II)

SECONDARY OBJECTIVES:

I. To determine the local and systemic toxicities associated with pulmonary suffusion. (Phase I) II. To determine whether suffusion improves metastatic control by suppressing progression of microscopic metastases to new lesions assessable by imaging (Phase I) III. To determine disease-free survival (DFS) in patients receiving pulmonary suffusion compared to historical controls, in patients with completely resected pulmonary metastases (unilateral and bilateral disease). (Phase II)

EXPLORATORY OBJECTIVES:

I. To evaluate the pulmonary suffusion-associated changes in local tumor microenvironment (TME) and potential of suffusion as an immune modulation enhancement. (Phase II) II. To determine overall survival (OS) in patients receiving pulmonary suffusion compared to historical controls, in patients with completely resected pulmonary metastases (unilateral and bilateral disease). (Phase II) III. To compare histology of tumor samples with previously resected specimens with attention to biomarkers of systemic immune recognition in patients eligible for repeat suffusion. (Phase II) IV. To obtain tumor and systemic immune biomarkers including cytokine activations for correlation with clinical responses. (Phase II) V. To correlate local control with biomarker for tissue effect from chemotherapy (including tissue levels of platinum, alkaline phosphatase [ALP]). (Phase II) VI. To correlate local disease control with tumor biomarker for metastasis (circulating [circ] ribonucleic acid [RNA], micro [mi]RNA). (Phase II)

OUTLINE:

Patients undergo pulmonary suffusion consisting of cisplatin via infusion. Patients then undergo metastasectomy. Patients found to have unresectable sarcoma may receive chemotherapy within 4-8 weeks of metastasectomy.

After completion of study treatment, patients are followed up for 3 months for one year and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Tumors metastatic to the lungs that are the focus of this protocol specifically:

  * Soft tissue sarcoma
  * Osteosarcoma
  * Colorectal carcinoma
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Hemoglobin > 8.0 g/L
* Granulocytes > 1,500 uL
* Platelets >= 100,000 uL
* Creatinine clearance >= 30 mL/min
* Clinically diagnosed resectable sarcoma lung metastases(while preregistration histologic or cytologic confirmation is desirable, this may not be required in clinical scenarios where a biopsy may not change the need to resect suspicious lung nodules or the biopsy itself poses a risk for tumor seeding. In such cases, the diagnosis will be supported by rapid pathologic evaluations intraoperatively before proceeding with Suffusion) Given the emergence of other acceptable options to destroy lung metastases such as SBRT or microwave ablation, a hybrid approach to eliminate all sites of disease will be permitted; however, supplemental approaches should be delayed, if possible, until after the 30 day post-suffusion endpoint
* Forced expiratory volume in 1 second (FEV1) >= 50% predicted
* Diffusion capacity of the lung for carbon monoxide (DLCO) >= 50% predicted
* Vital capacity (VC) >= 50% predicted
* Ambulatory and resting oxygen (O2) saturation > 88%
* Six minute walk >= 50 % of the expected distance
* Surgeon affirmation that suffusion is technically feasible
* Borg Dyspnea scale (modified) < 5
* Control of the primary tumor as determined by clinical assessment per standard of care; may include stable tumor status of primary tumor and other metastases, in the clinical judgement of the PI/Physician.
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Allergy, intolerance, or other serious reaction to chemotherapy drugs that may be used in the procedure
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Pulmonary metastases unable to be completely resected or ablated based on pre-registration review of imaging by a thoracic surgeon or proceduralist.
* Any additional condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive study drug or the suffusion technique, may include uncontrolled intercurrent illness and other conditions that, in the judgement of the PI/Physician, would limit compliance with the study requirements and have safety concerns
* Received an investigational agent within 30 days prior to enrollment
* Severe peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2020-07-16 (Actual); Primary Completion 2029-05-25 (Estimated); Study Completion 2030-05-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of local toxicities (Phase I) | Up to 2 years
  Dose limiting toxicities (DLTs) will be defined based on the rate of drug-related grade 3-5 adverse events. These will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.
Recommended phase II dose (Phase I) | Up to 5 years
Local recurrence (Phase II) | From resection until local recurrence in the suffused lung or last clinic follow-up, assessed up to 2 years
  Will be treated as bivariate time-to-event data. Freedom from local recurrence will be summarized using standard Kaplan-Meier methods and the 2-year local recurrence-free rate will be estimated with a 90% confidence interval calculated using Greenwood's formula.

SECONDARY OUTCOMES:
Incidence of local and systemic toxicities (Phase I) | Up to 5 years
  Assessed using the NCI CTCAE v5.0.
Disease-free survival (Phase II) | From suffusion until recurrence (local or distant), death due to or related to disease, or last follow-up, assessed up to 2 years
  Will be summarized using standard Kaplan-Meier methods, where estimates of the median survival and 2-year survival rates will be obtained with 90% confidence intervals.
Incidence of local and systemic toxicities (Phase II) | Up to 5 years
  Assessed using the NCI CTCAE v5.0. Will be summarized by grade within each arm using frequencies and relative frequencies.
Local recurrence within the treated (suffusion) and untreated lungs for patients with bilateral disease (Phase II) | At 2 years
  Will be compared between the suffused and non-suffused lungs using McNemar?s test. A 90% confidence interval about the difference in local recurrence rates will also be obtained.

OTHER OUTCOMES:
Lung injury (% reduction of spirometry and differential reduction by quantitative perfusion scan) (Phase II) | Up to 5 years
  The association between lung injury and response and survival outcomes will be evaluated using logistic and Cox regression models.
Immune markers (Phase II) | Up to 5 years
  Will be correlated to primary endpoints. The cytokine activation, tumor, immune, and stress related biomarkers will be summarized using the appropriate descriptive statistics. The association between overall response and the biomarkers will be evaluated using logistic regression models. The association between time-to-event outcomes (freedom from recurrence and survival) and the biomarkers will be evaluated using Cox regression models. All model assumptions will be verified graphically and fit using Firth's method.
Overall survival (Phase II) | Up to 5 years
  Will be compared to historical controls. Will be summarized using standard Kaplan-Meier methods, where estimates of the median survival and 2-year survival rates will be obtained with 90% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Todd L Demmy, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States